CLINICAL TRIAL: NCT00950534
Title: A Randomised, Multicentre, Open-Label, Parallel-Group, 24-Week Phase IV Study Comparing the Effectiveness and Safety of Two Approaches to the Management of Type 2 Diabetes Mellitus in Australian Primary Care: General Practitioner Initiation of Insulin Glargine Versus the Usual Standard of Care
Brief Title: Effectiveness and Safety of Two Approaches to the Management of Type 2 Diabetes Mellitus in Australian Primary Care
Acronym: RELIANCE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: due to poor recruitment
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_L_04264
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Hypoglycemic Agents

ARMS (2):
- General Practitioner initiation with insulin glargine (Experimental): Patients will be prescribed insulin glargine by their Investigator and they will be taught how to administer insulin glargine according to Australian guidelines. Patients will be treated for 24 weeks.
  Interventions: Drug: INSULIN GLARGINE (HOE901)
- Usual standard of care (Active Comparator): Patients will be treated by their Investigator with the usual standard of care for 24 weeks (e.g., OAD dose titration, addition of a second or third OAD, or referral to an endocrinologist)
  Interventions: Drug: Oral Anti Diabetics (OAD)

INTERVENTIONS:
Drug: INSULIN GLARGINE (HOE901) — The dose of insulin glargine will be titrated toward a fasting plasma glucose (FPG) target of 5.5 mmol/L. Treatment with oral antidiabetic drugs (OADs) prescribed before study entry may continue (except Sitagliptin, Acarbose, Rosiglitazone)
  Arms: General Practitioner initiation with insulin glargine
Drug: Oral Anti Diabetics (OAD) — Patients treated with the usual standard of care (OAD dose titration, addition of a second or third OAD or referral to an endocrinologist) until optimal doses are reached to maintain a FPG of 5.5 mmol/L
  Arms: Usual standard of care

SUMMARY:
The primary objective is to demonstrate the improvement in glycosylated haemoglobin (HbA1c) levels after general practitioner (GP) initiation and management of type 2 diabetes mellitus (T2DM) with insulin glargine compared with their usual clinical practice.

The secondary objective is to demonstrate the importance of GP initiation of insulin glargine for the treatment of T2DM.

ELIGIBILITY:
Inclusion criteria:

* Diagnosed with type 2 Diabetes Mellitus (T2DM)
* HbA1c > or = 7.5%, or HbA1c < or = 10%
* Continuous oral antidiabetic (OAD) treatment for more or equal than three months before randomisation with stable daily doses of one or more OADs (if on two or more OADs, one must be less or equal than half maximum tolerated dose)
* Willing and able to perform blood glucose monitoring using a blood glucose meter
* Willing and able to keep a daily patient diary
* Willing and able to provide written informed consent before enrolment in the study

Exclusion criteria:

* Type 1 diabetes mellitus
* Body mass index (BMI) > 45 kg/m²
* Works night shifts
* History of ketoacidosis or hyperosmolar hyperglycaemic state
* History of stroke, myocardial infarction, angina pectoris, coronary artery bypass graft or percutaneous transluminal coronary angioplasty within the previous 12 months
* History of congestive heart failure
* Hypoglycaemia unawareness
* Have had more than one episode of hypoglycaemia (per protocol definition) within 24 weeks before screening
* Impaired renal function defined as, but not limited to, serum creatinine > or = 1.5 mg/dL (133 µmol/L) males or > or = 1.4 mg/dL (124 µmol/L) females
* Active liver disease (alanine transaminase (ALT) greater than two times the upper limit of the reference range, as defined by the local laboratory)
* Have any condition (including known substance or alcohol abuse or psychiatric disorder) that precludes the patient from following and completing the study protocol
* Had a blood transfusion or severe blood loss within the 3 months before screening, or have known haemoglobinopathy, haemolytic anaemia or sickle cell anaemia
* Current or previous use of insulin
* Known hypersensitivity / intolerance to insulin glargine or any of its excipients
* Have taken exenatide in the six weeks before screening or for a total of 30 days or more in the 24 weeks before screening
* Currently receiving treatment with non-selective -blockers
* Currently receiving chronic (longer than two weeks) systemic glucocorticoid therapy (excluding topical or inhaled preparations) or have received such therapy within the four weeks preceding the screening visit
* Currently undergoing therapy or planned radiological examinations requiring the administration of contrasting agents for malignancy (other than non-metastatic / early stage basal cell or squamous cell carcinoma).
* Currently participating in another investigational study or recent study participation ending < 30 days before screening
* Female patients who are pregnant or breastfeeding
* Female patients of childbearing potential (i.e., ovulating, pre-menopausal, not surgically sterile) must be willing to agree to use a medically accepted contraceptive regimen for the duration of the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The percentage of patients achieving glycosylated haemoglobin (HbA1c) levels < or = 7.0% | From week 0 to week 24

SECONDARY OUTCOMES:
Time required to reach the target HbA1c level of < or = 7% | From week 0 to week 24
The percentage of patients achieving two consecutive on treatment HbA1c measurements of < or = 7.0% | From week 0 to week 24
Decrease in mean HbA1c level | At week 24
Decrease in mean Fasting Plasma Glucose (FPG) | At week 24
Mean change in body weight | At week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Macquarie Park, Australia